CLINICAL TRIAL: NCT03504358
Title: A New Prognostic Scoring System for Spontaneous Ruptured Hepatocellular Carcinoma: A Retrospective Study
Brief Title: A New Prognostic Scoring System for Spontaneous Ruptured Hepatocellular
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoping Chen, Professor, Huazhong University of Science and Technology
Other Study IDs: Zhupeng002
Record Dates: First submitted 2018-04-04; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Rupture, Spontaneous
Keywords: surgery; scoring system; hepatocellular carcinoma; homogeneity and discriminatory ability; survival
MeSH Terms: conditions — Rupture, Spontaneous; Carcinoma, Hepatocellular | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Analysis before liver resection: Multivariate analysis of predictive factors associated with survival
  Interventions: Procedure: Liver resection
- Different risk group: Low-risk group, moderate-risk group, high-risk group
  Interventions: Procedure: Liver resection
- Model comparison: Comparison of models in predicting survival
  Interventions: Procedure: Liver resection

INTERVENTIONS:
Procedure: Liver resection — Partial hepatectomy comprised single or multiple hepatic resections aiming at excising all visible malignant tissue.

SUMMARY:
Develop a new scoring system for HCC patients with tumor rupture.

DETAILED DESCRIPTION:
There has been no special prognostic scoring system for HCC patients with tumor rupture in the literature. In this work, we obtained all survival risk factors of ruptured HCC patients who underwent partial hepatectomy using multivariable Cox regression analysis. Furthermore, we develop and validate a new postoperative scoring system for patients with spontaneous HCC rupture based on the these results.

ELIGIBILITY:
Inclusion Criteria:

* Received partial hepatectomy; with Child A or B liver function.

Exclusion Criteria:

* Without complete data；loss of follow-up; had reveived repeated transcatheter arterial chemoembolization before rupture; received non-radical resection.

Ages: 15 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Ten year HCC rupture patients who received partial hepatectomy at Tongji Hospital of the Huazhong University of Science and Technology
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years
  Overall survival after partial hepatectomy

SECONDARY OUTCOMES:
Disease-free survival | 3 years
  Recurrence-free survival after partial hepatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Bi-xiang Zhang, Prof, PHD, Study Chair — Huazhong University of Science and Technology